CLINICAL TRIAL: NCT05076383
Title: The Effect of Motor Re-Learning Program on Balance, Mobility and Performance of Activities of Daily Living Among Post-Stroke Patients: A Randomized Controlled Trial
Brief Title: The Effect of Motor Learning on Balance, Mobility and Performance of Activities of Daily Living Among Post-Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Parc de Salut Mar (Other)
Responsible Party: Principal Investigator, Amer Ghrouz, Principal Investigator, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021/9986/I
Record Dates: First submitted 2021-09-22; First posted 2021-10-13 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Stroke
Keywords: Rehabilitation; Motor learning; Balance; Mobility
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motor relearning program (MRP) (Experimental)
  Interventions: Other: Study Group (Motor relearning program)
- Conventional physical therapy program (CPT) (Active Comparator)
  Interventions: Other: Control Group (Conventional physical therapy program)

INTERVENTIONS:
Other: Study Group (Motor relearning program) — Task-specific training based on motor relearning program will be performed for 8 weeks (3 sessions per week; 1 hr. per session; total 24 sessions). Each training session will consist of five training tasks: (1) bed mobility and sitting up over the side of the bed; (2) balanced sitting; (3) standing up and sitting down; (4) balanced standing; and (5) practice of walking.
  Arms: Motor relearning program (MRP)
Other: Control Group (Conventional physical therapy program) — The conventional physical therapy program (CPT) exercises will be performed following a standard stroke rehabilitation program for 8 weeks (3 sessions per week; 1 hr. per session; total 24 sessions). Each CPT rehabilitation session will include the following exercises: (1) passive and active-assisted range of motion; (2) stretching; (3) strengthening exercises; (4) balance exercises; and (5) walking.
  Arms: Conventional physical therapy program (CPT)

SUMMARY:
The primary objective of this study is to assess - through a randomized controlled trial - the effectiveness and long-term improvement of motor relearning program on balance, mobility and performance of activities of daily living among post-stroke patients. In this two-armed randomized controlled clinical trial, a total of 66 sub-acute stroke patients who meet the trial criteria will be recruited. The patients will randomly receive task-specific training based on a motor relearning program (MRP) or a conventional physical therapy program (CPT). Twenty-four rehabilitation sessions will be conducted for eight weeks. Both interventions will be followed by analysis of patients' balance, gait and performance of activates of daily living at two time period; post-intervention and follow-up after 3-months, using clinical outcome measures and instrumental analysis of balance and gait.

ELIGIBILITY:
Inclusion Criteria:

* First-ever subacute (1-6 months) stroke patients;
* Able to give informed consent;
* Patients with hemiparesis: muscle power of 2-4 on Medical Research Council-MRC Muscle Scale in the affected upper and lower limbs;
* Able to stand independently for at least one minute;
* Can ambulate 25 feet/10 meter (with or without assistive device).

Exclusion Criteria:

* Post-stroke patients with major cognitive deficits (Montreal Cognitive Assessment- MoCA score ≥ 20) and/or communication impairments that don't allow patients to follow directions (i.e., deafness, aphasia, etc.);
* Patients who are receiving other related therapy through the study, which may affect efficacy of this study;
* Any medical contraindications to start rehabilitation;
* History of disability related to neurological deficits other than stroke.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale (BBS) | The BBS will be used to assess the changes from the baseline balance at 8 weeks (post-intervention) as well as at 3-months after intervention (3-months follow-up).
Timed Up and Go Test (TUG) | The TUG will be used to evaluate the changes from baseline functional mobility at 8 weeks (post-intervention) as well as at 3-months after intervention (3-months follow-up).
10-meter Walk Test (10mWT) | The 10mWT will be used to assess the changes from the baseline walking speed (meters per second) at 8 weeks (post-intervention) as well as at 3-months after intervention (3-months follow-up).
Barthel Index (BI) | The BI will be used to measure the changes from baseline functional independency at 8 weeks (post-intervention) as well as at 3-months after intervention (3-months follow-up).
Instrumental analysis of balance | NedSVE/IBV® system will be used to assess the changes from baseline balance and postural control at 8 weeks (post-intervention) as well as at 3-months after intervention (3-months follow-up).
  The balance and postural control will be assessed using the computerized posturography - NedSVE/IBV® platform.
Instrumental analysis of gait | NedAMH/IBV® system will be used to assess the changes from baseline gait parameters at 8 weeks (post-intervention) as well as at 3-months after intervention (3-months follow-up).
  The gait will be assessed using the NedAMH/IBV® system, a software application for the biomechanical gait assessment, based on the use of a Dinascan/IBV P600 dynamometric platform.

CONTACTS AND LOCATIONS:
Overall Officials: Amer Ghrouz, PhD Student, Principal Investigator — Physical Medicine and Rehabilitation, Centre Fòrum, Parc de Salut Mar, Barcelona, Spain; Esther Duarte, MD, PhD, Study Director — Physical Medicine and Rehabilitation, Hospitals del Mar i l'Esperança, Parc de Salut Mar, Barcelona, Spain
Locations (1):
- Centre Fòrum, Parc de Salut Mar, Barcelona, Spain

REFERENCES:
- [Derived] Ghrouz A, Marco E, Munoz-Redondo E, Boza R, Ramirez-Fuentes C, Duarte E. The effect of motor relearning on balance, mobility and performance of activities of daily living among post-stroke patients: Study protocol for a randomised controlled trial. Eur Stroke J. 2022 Mar;7(1):76-84. doi: 10.1177/23969873211061027. Epub 2022 Feb 11. PMID 35300258